CLINICAL TRIAL: NCT01724957
Title: Fractional Flow Reserve Versus Intracoronary ECG for Detection of Post Stenting Ischemia in Side Branch Territory in coronAry Bifurcation Lesions
Brief Title: FFR vs. icECG in Coronary Bifurcations
Acronym: FIESTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University National Heart Hospital (Other)
Responsible Party: Principal Investigator, Dobrin Vassilev, Dobrin Vassilev MD, PhD, University National Heart Hospital
Other Study IDs: 20120109-05
Record Dates: First submitted 2012-11-05; First posted 2012-11-12 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease
Keywords: Fractional flow reserve,; coronary bifurcation stenosis,; intracoronary ECG,; coronary stent; Coronary bifurcation lesions; icECG
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with coronary bifurcation lesions: Only one group will be studied. The patient will be a slef-reference.
  Interventions: Procedure: Intracoronary ECG

INTERVENTIONS:
Procedure: Intracoronary ECG — Recording of icECG from the tip of PCI guidewire. The wire end is connected through alligator clips to V-lead from surface ECG

SUMMARY:
The study hypothesis: it is possible to use icECG recorded from regular PCI wire to predict significance of SB ostial stenosis after main vessel stenting in coronary bifurcation lesions.

DETAILED DESCRIPTION:
The coronary bifurcation lesions pose a therapeutic problem with high rates of periprocedural complications, higher rates of in-stent restenosis and stent thrombosis. These are lesions where stenting is not superior in comparison to balloon angioplasty in regard to side branch. It was demonstrated many times, in literature and in daily practice, that angiographically high grade ostial side branch stenosis is not flow limiting and do not cause ischemia, therefore do not require treatment. From the other side, our own data with MRI before and after bifurcation PCI demonstrated that occurrence of angiographic stenosis more than 70% in diameter is associated with periprocedural myonecrosis in the region of side branch. This fact puts a very important question about the mechanisms of this myonecrosis. If the jailed side branch has no significant flow limiting stenosis, but there is some degree of residual ischemia, which after some period of persistence could lead to myonecrosis, will mean that more aggressive treatment of ostial stenosis is needed. It is interesting that the strategy of treatment is very important, because techniques with second stent implantation (with primary purpose to limit SB ischemia) are associated with higher grade of troponin increase. Of course this is association and not causality, despite that in randomized study (NORDIC I) it was confirmed also.

It is without explanation the fact of rare occurrence of significant (flow limiting, FFR <.75) stenosis appearance (less than 40% in side branches with ostial stenosis more than 75%) and almost 50% periprocedural myonecrosis detected in the side branch areas. One working hypothesis is that stent implantation and related episode of ischemia induces prolonged vasospasm, resulting in prolonged ischemia. Thus, the ostial stenosis could be non-significant as estimated and registered by FFR, but on microcirculatory lever ischemia could persist is small areas for which available flow is not sufficient despite that global regional flow is deemed sufficient. It is also possible that those patients have not enough recruitable collaterals. It is also possible that both factors act together.

Although FFR is useful for assessing the degree of ischemia caused by a coronary lesion, it cannot give information as to whether this ischemia may be clinically significant or not, i.e. whether the ischemia affects a large territory. Therefore, it can be implicated that FFR may not be useful in predicting clinically meaningful ischemia in a specific side branch vessel.

The intracoronary electrocardiography (i.c. ECG) is a very sensitive method for ischemia detection. The i.c. ECG reacts earlier on ischemia; the changes are much more prominent and easy to register. The wire tip could be positioned directly in different regions and thus to "map" regional ischemia. In most of the studies and from our own observations became evident that when surface ECG do not react the i.c. ECG demonstrates significant changes in ST-segment and QRS complex. Moreover, the registration of i.c. ECG is very cheap and needs only an adapter connecting coronary wire end and ECG. An i.c. ECG also can differentiate residual ischemic changes in distal main vessel and side branch as sources of prolonged ischemia, respectively - source of periprocedural myonecrosis.

The objective of this study is to evaluate concordance between icECG findings and FFR findings after stenting main vessel.

ELIGIBILITY:
Inclusion Criteria:

* Subject at least 18 years of age.
* Subject able to verbally confirm understandings of risks, benefits of receiving PCI for true bifurcation lesions, and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
* Target main branch lesion(s) located in a native coronary artery with diameter of ≥ 2.5 mm and ≤ 4.5 mm. Target side branch lesion(s) located in a native coronary artery with diameter of ≥ 2.0 mm.
* Target lesion(s) amenable for PCI with balloon angioplasty of the side branch.

Exclusion Criteria:

* Subjects with significant ST-T change (≥ 1mm).
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Subjects who refuse to give informed consent.
* Subjects with the following angiographic characteristics: left main coronary artery stenosis, total occlusion before occurrence of SB, lesion of interest located at infarct-related artery.
* Subjects with LVEF < 30%.
* Subjects with moderate or severe degree valvular heart disease or primary cardiomyopathy.
* LBBB, RBBB, atrial fibrillation/flutter with no identifiable isoelectric line.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Significant, >50% diameter stenosis artery scheduled for stent insertion at the main vessel (Medina types: 1xx, x1x, 11x);
  * Side branch vessel at least 2.0mm
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-12 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Side branch region ischemia duration | Percutaneous coronary intervention procedure time (up to 4h)
  FFR<0.80 at the SB ostium after stenting main vessel in coronary bifurcation lesion; icECG ST-segment elevation >2.0mm; T-wave inversion >3mm; ST-segment depression >2mm, not observed at the beginning of procedure

SECONDARY OUTCOMES:
Target lesion revascularization | 12 months
  Any revascularization at the territory of previously implanted stent.
Number of patients not alive | 12 month
Myocardial infarction after hospital discharge | 12 months
  MI according to universal definition of MI - CK-MB > 2xULN +/- symptoms +/- surface ECG changes in at least 2 leads
New onset angina or heart failure symptoms | 12 months
  New onset angina symptoms of at least CCS class II; New onset dyspnea at exertion or at rest

OTHER OUTCOMES:
Periprocedural myonecrosis - extent of post PCI enzyme elevation | 48h
  Troponin I elevation 1-3; 3-5; >5 x ULN Creatin phospho kinase MB fraction elevation 1-3; 3-5; >5 x ULN

CONTACTS AND LOCATIONS:
Locations (2):
- Indiana-Purdue University, Indianapolis, Indiana, United States
- National Heart Hospital, Sofia, Bulgaria